CLINICAL TRIAL: NCT06888102
Title: IIT2023-10-Posadas-PC-Net : A Platform Study of Epigenetic Therapy Before Prostatectomy in Men With Prostate Cancer
Brief Title: A Platform Study of Epigenetic Therapy Before Prostatectomy in Men With Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Edwin Posadas, MD (Other)
Responsible Party: Sponsor-Investigator, Edwin Posadas, MD, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-10-Posadas-PC-NET
Record Dates: First submitted 2024-10-11; First posted 2025-03-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: High-risk Prostate Cancer
Keywords: Epigenetic Therapy; PD-L1; radical prostatectomy

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized platform protocol opening multiple modules, not running concurrently. Each module will enroll 20 patients. Module A will use open-label azacitidine in the neoadjuvant setting for patients with a diagnosis of prostate cancer undergoing radical prostatectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Epigenetic Therapy (Experimental)
  Interventions: Drug: Neoadjuvant Epigenetic Therapy

INTERVENTIONS:
Drug: Neoadjuvant Epigenetic Therapy — Participants will be assigned to receive one of the study interventions and will be monitored for safety and response. The duration of epigenetic therapy will be dependent on the treatment administered and will continue for the duration described in the cohort appendix for each respective combination, unless the participant: is no longer clinically benefiting (NLCB, as evidenced by symptomatic or radiographic disease progression and/or clinical deterioration); experiences any toxicity meeting specified discontinuation criteria (as described in the cohort appendix for each respective combination) or unacceptable toxicity in the best clinical discretion of the treating physician (i.e., Investigator discretion); reaches the maximum duration of study intervention; or withdraws consent.

SUMMARY:
This is an open-label, non-randomized, exploratory platform protocol designed to assess the safety and antitumor activity of epigenetic therapies in participants with localized prostate cancer who are undergoing radical prostatectomy. The epigenetic therapy is intended to increase the sensitivity of the underlying tumor to the patient's immune system. The platform study will evaluate safety, biomarkers, and clinical activity of an epigenetic therapy. The particular details relevant to each module within this platform study will be provided as appendices to the core protocol.

DETAILED DESCRIPTION:
The study lead investigators will modify and/or add new therapies to the protocol as data emerge from this and other trials. Participants must provide consent for archival biopsy tissue prior to surgery for prostate cancer and must consent to allowing for use of their surgical specimens from biopsy and prostatectomy for biomarker characterization. Given the absence of data in this setting, this pilot proposes this experience with up to 4 weeks of epigenetic agents at doses known to be clinically safe and effective at inducing clinical activity.

Participants will be assigned to receive one of the study interventions and will be monitored for safety and response. The duration of epigenetic therapy will be dependent on the treatment administered and will continue for the duration described in the cohort appendix for each respective combination, unless the participant: is no longer clinically benefiting (NLCB, as evidenced by symptomatic or radiographic disease progression and/or clinical deterioration); experiences any toxicity meeting specified discontinuation criteria (as described in the cohort appendix for each respective combination) or unacceptable toxicity in the best clinical discretion of the treating physician (i.e., Investigator discretion); reaches the maximum duration of study intervention; or withdraws consent.

ELIGIBILITY:
Inclusion Criteria

* Men electing to undergo radical prostatectomy with preoperative tissue available.
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate organ function defined by:

  * AST and ALT < 2.5 x ULN
  * Total bilirubin < 1.5 x ULN
  * Platelets > 90 x 1000/μL
  * Hemoglobin (Hgb) > 8.5 g/dL
  * Serum Creatinine (Cr) <1.5 x ULN or eGFR > 30 mL/min
* People with partners of childbearing potential in circumstances that may result in the pregnancy, must have had a successful vasectomy (with medically confirmed lack of sperm that are alive) OR must either practice complete abstinence or agree to use adequate contraception (latex or synthetic condom during sexual contact with a female of childbearing potential) from the start of study treatment until 3 months following last dose of study intervention. Subjects should not donate sperm on study, during interruptions in treatment and for 3 months following completion of study drug treatment.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria

* Active intercurrent illness or malignancy requiring therapy outside of prostate cancer.
* Other anti-cancer therapy (chemotherapy, hormonal therapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization)
* Currently participating in a study using an investigational, medicinal anti-cancer agent within 4 weeks prior to first dose of epigenetic therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Safety of Using Epigentic Therapy | 2 Years
  Safety and tolerability using CTCAE version 5.0. To assess the safety, toxicity, and feasibility of using epigenetic therapy in the neoadjuvant setting for men undergoing radical prostatectomy (RP). Defined by the number of patients who demonstrate treatment related AEs, defined as grade 3 or 4, or grade 2 that causes a dose interruption.
Toxicity of Using Epigentic Therapy | 2 Years
  Safety and tolerability using CTCAE version 5.0. To assess the safety, toxicity, and feasibility of using epigenetic therapy in the neoadjuvant setting for men undergoing radical prostatectomy (RP). Defined by the number of patients that undergo radical prostatectomy without delay due to epigenetic therapy.
Feasibility - % of Patients Able to Undergo Surgery | 2 Years
  Feasibility - Percentage of patients able to undergo surgery. To assess the feasibility of measuring changes in gene expression (in radical prostatectomy [RP] tissue) induced by epigenetic therapy at conventional doses (defined by ongoing clinical work focusing on doses within the recommended dose and schedule per the manufacturer where safety has been defined) with a focus on Interferon Stimulated Genes
Feasibility - % of patients with grade 3/4 AEs related | 2 Years
  Feasibility - Percentage of patients with grade 3/4 adverse events related to epigenetic therapy. To assess the feasibility of measuring changes in gene expression (in radical prostatectomy [RP] tissue) induced by epigenetic therapy at conventional doses (defined by ongoing clinical work focusing on doses within the recommended dose and schedule per the manufacturer where safety has been defined) with a focus on Interferon Stimulated Genes
Feasibility - % of patients with evaluable tissue specimens | 2 Years
  Feasibility - Percentage of patients with evaluable tissue specimens following epigenetic therapy. To assess the feasibility of measuring changes in gene expression (in radical prostatectomy [RP] tissue) induced by epigenetic therapy at conventional doses (defined by ongoing clinical work focusing on doses within the recommended dose and schedule per the manufacturer where safety has been defined) with a focus on Interferon Stimulated Genes. The evaluability of tissue specimens would be defined as the number of subjects that completed epigenetic therapy and underwent RP and undergo any of the correlative studies using tissue or blood.

SECONDARY OUTCOMES:
Progression Free Survival | 7 Years
  To estimate the biochemical progression free survival in men treated with epigenetic therapy prior to prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Cancer at SOCC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No